CLINICAL TRIAL: NCT04024995
Title: Revision of Antifungal Strategies Definitions for Invasive Fungal Infections (Proven/Probable/Possible) in Patients With Hematological Malignancies (REDEFI-SEIFEM)
Brief Title: Revision of Antifungal Strategies Definitions for Invasive Fungal Infections in Hematological Malignancies
Status: Completed | Type: Observational
Sponsor: Sorveglianza Epidemiologica Infezioni Fungine Emopatie Maligne (Other)
Responsible Party: Principal Investigator, LIVIO PAGANO, Associate professor, Sorveglianza Epidemiologica Infezioni Fungine Emopatie Maligne
Other Study IDs: REDEFI-SEIFEM
Record Dates: First submitted 2019-02-26; First posted 2019-07-18 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Invasive Fungal Infections
Keywords: Invasive Fungal Infections; EORTC/MSG criteria
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to evaluate invasive fungal infections (IFI) according to clinicians' opinion vs the opinion of an independent board of experts. The primary output of this study is the evaluation of inter-raters agreement. Secondary objectives are: evaluation of IFI incidence; description of clinical and laboratory features; frequencies of different antifungal treatments; description of outcome; impact on the treatment of underlying hematological malignancy. This is a multicenter, non-interventional observational, prospective study. The duration of the study will be 18 months. The study will recruit all consecutive eligible patients in each participating center, during a period of 6 months until at least 600 patients with acute myeloid leukemia are registered, that represented the highest risk category. Other disease types that fulfill the eligibility criteria in the participating centers during the same period will also be recruited in the study.

The clinical, microbiological, diagnostic and therapeutic procedures operated on these patients will be collected.

An eCRF will be compiled for all patients:

T0: at the start of antifungal treatment, information will be collected regarding hematological malignancy, status of the disease at onset of infection and phase of treatment, last chemotherapy regimen, comorbidities and risk factors; previous IFI, neutropenia, antifungal and antibiotic prophylaxis and the kind of IFI clinicians retain the patient suffer (possible/probable/proven) and the kind of antifungal treatment started (empiric/pre-emptive/target); diagnostic work-up done, positive microbiology and biomarkers, positive radiological findings; antifungal treatment.

T1: at 30-40 days (or before if the patient unfortunately died) a second form must be completed with information regarding any changes in/additional diagnostic work-up done, positive microbiology and biomarkers, positive radiological findings; any changes in antifungal treatment; outcome.

At that time, the local physician must state any revision of his diagnostic classification between the moment in which antifungal treatment was started and the moment of evaluation of the outcome in order to estimate the differences regarding the level of evidence of diagnosis and treatment of IFI during time.

Each case will be examined blinded by 2 different experts, who will review all records based on the existing guidelines, their own experience and the information that was known at the two time points, which may confirm or not the decision of local physician.

The sample size will be driven by the AML patients (approximately 60-70% of the patients). Sample will be described in its clinical and demographic features via descriptive statistics. Quantitative variables will be summarized with the following measures: minimum, maximum, range, mean and standard deviation. Qualitative variables will be represented by frequencies tables.

DETAILED DESCRIPTION:
Primary objective The primary objective of this study is to evaluate IFI according to clinicians' opinion vs the opinion of an independent board of experts. The independent panel, confirming or not the decision of local physician, will review all cases (blind central review). The primary output of this study is the evaluation of inter-raters agreement.

Secondary objectives:

Evaluation of IFI incidence Description of clinical and laboratory features Frequencies of different antifungal treatments Description of outcome Impact on the treatment of underlying hematological malignancy

Study design This is a multicenter, non-interventional observational, prospective study.

The duration of the study will be 18 months. The schedule for the study will be the following:

Observation and data collection: 6 months Revision board: 6 months Data elaboration and paper: 6 months

Materials and methods The study will recruit all consecutive eligible patients in each participating center, during a period of 6 months until at least 600 AML patients are registered, that represented the highest risk category of patients for IFI. Other disease types that fulfill the eligibility criteria in the participating centers during the same period will also be recruited in the study.

We do not expect that diagnostic work-up would significantly vary among the participating centers. Minimal diagnostic work up must include:

Blood cultures for fungal infection; Chest High Resolution CT-scan; Serum galactomannan; Sinus CT-scan (if indicated); Bronchoalveolar lavage (if indicated);

Centers participating to the study will be selected on the basis of a questionnaire that evaluate their availability to participate to the survey (see Appendix 1).

The clinical, microbiological, diagnostic and therapeutic procedures operated on these patients will be collected.

An electronic CRF will be compiled for all patients at two different time points: T0 and T1.

T0: at the start of antifungal treatment (study entry), information will be collected regarding:

Hematological malignancy, status of the disease at onset of infection and phase of treatment, last chemotherapy regimen, comorbidities and risk factors (previous allogeneic stem cell transplantation); Previous IFI, neutropenia, antifungal and antibiotic prophylaxis: the local physicians must define the kind of IFI they retain the patient suffer (possible/probable/proven) and the kind of antifungal treatment started (empiric/pre-emptive/target); Diagnostic work-up done, positive microbiology and biomarkers, positive radiological findings; Antifungal treatment.

T1: at 30-40 days (or before if the patient unfortunately died) a second form must be completed with information regarding:

any changes in/additional diagnostic work-up done, positive microbiology and biomarkers, positive radiological findings; any changes in antifungal treatment; outcome. At that time, the local physician must state any revision of his diagnostic classification between the moment in which antifungal treatment was started and the moment of evaluation of the outcome (30 days) in order to estimate the differences regarding the level of evidence of diagnosis and treatment of IFI during time.

Independent central review board The experts (each case will be examined blinded by 2 different experts). The experts will review all records based on the existing guidelines, their own experience and based on the information that was known at the two time points, which may confirm or not the decision of local physician.

Statistical considerations Sample size dimension The sample size will be driven by the AML patients (approximately 60-70% of the patients): Statistical analysis Sample will be described in its clinical and demographic features via descriptive statistics. Quantitative variables will be summarized with the following measures: minimum, maximum, range, mean and standard deviation. Qualitative variables will be represented by frequencies tables (absolute and percentage) The primary object of the study will be achieved evaluating Fleiss' Kappa. Secondary objectives will be using descriptive statistics techniques (already described above) recruit all eligible patients during a period of 6 months until at least 600 AML patients are recruited.

ELIGIBILITY:
Inclusion Criteria:

* All patients with hematologic malignancies at any stage of the disease (acute myeloid leukemia, acute lymphoblastic leukemia, multiple myeloma, myelodysplastic syndromes, chronic lymphocytic leukemia, high and low grade non Hodgkin lymphoma, chronic myeloprolipherative disorders, Hodgkin lymphoma);
* Only inpatients will be eligible;
* Patient that start IV antifungal treatment (irrespective of previous prophylaxis);
* Informed consent signed.

Exclusion Criteria:

* Patients with previous or undergoing allogeneic or autologous transplant will be excluded from the study, due to different clinical profiles and risk factors;
* Patients treated, after prophylaxis with oral antifungals
* Patients treated in outpatient clinic or Day hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will recruit all consecutive eligible patients in each participating center, during a period of 6 months until at least 600 AML patients are registered, that represented the highest risk category of patients for IFI. Other disease types that fulfill the eligibility criteria in the participating centers during the same period will also be recruited in the study.
Sampling Method: Non-Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of diagnosis Agreement in proven/probable/possible IFI in real life using EORTC/MSG Criteria | 30 days
  Rate of diagnosis agreement in proven/probable/possible IFI between local physician in real life and indipendent board of experts according to EORTC/MSG Criteria

SECONDARY OUTCOMES:
Evaluation of incidence of invasive fungal infections | 6 months
  Evaluation of incidence of IFI among hematological patients
Attributable and all-cause mortality of patients with invasive fungal infections | 30 days
  Description of attributable and all-cause mortality of hematological patients with IFI

CONTACTS AND LOCATIONS:
Overall Officials: Livio Pagano, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli IRCCS-UCSC
Locations (14):
- Italy (14):
  - Azienda Ospedaliera Universitaria S. Orsola Malpighi, Bologna
  - ASST-Spedali Civili, Brescia
  - AOUC Carreggi, Florence
  - AOU Policlinico Federico II, Napoli
  - Azienda Ospedaliera di Perugia, Perugia
  - Azienda Ospedaliera San Camillo Forlanini, Rome
  - Fondazione Policlinico A. Gemelli IRCCS, Rome
  - Istituto Nazionale Tumori Regina Elena IFO, Rome
  - Ospedale Infantile Regina Margherita, Torino
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine
  - Osp. di Circolo-Fondazione Macchi, Varese
  - AOUI Verona, Verona
  - Ospedale Donna Bambino, Verona
  - Ospedale San Bortolo- AULSS 8 Berica, Vicenza

REFERENCES:
- [Background] De Pauw B, Walsh TJ, Donnelly JP, Stevens DA, Edwards JE, Calandra T, Pappas PG, Maertens J, Lortholary O, Kauffman CA, Denning DW, Patterson TF, Maschmeyer G, Bille J, Dismukes WE, Herbrecht R, Hope WW, Kibbler CC, Kullberg BJ, Marr KA, Munoz P, Odds FC, Perfect JR, Restrepo A, Ruhnke M, Segal BH, Sobel JD, Sorrell TC, Viscoli C, Wingard JR, Zaoutis T, Bennett JE; European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group; National Institute of Allergy and Infectious Diseases Mycoses Study Group (EORTC/MSG) Consensus Group. Revised definitions of invasive fungal disease from the European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group and the National Institute of Allergy and Infectious Diseases Mycoses Study Group (EORTC/MSG) Consensus Group. Clin Infect Dis. 2008 Jun 15;46(12):1813-21. doi: 10.1086/588660. PMID 18462102
- [Background] Mercier T, Maertens J. Clinical considerations in the early treatment of invasive mould infections and disease. J Antimicrob Chemother. 2017 Mar 1;72(suppl_1):i29-i38. doi: 10.1093/jac/dkx031. PMID 28355465
- [Background] Maccioni F, Vetere S, De Felice C, Al Ansari N, Micozzi A, Gentile G, Foa R, Girmenia C. Pulmonary fungal infections in patients with acute myeloid leukaemia: is it the time to revise the radiological diagnostic criteria? Mycoses. 2016 Jun;59(6):357-64. doi: 10.1111/myc.12480. Epub 2016 Feb 11. PMID 26865204
- [Background] Cornely OA, Maertens J, Winston DJ, Perfect J, Ullmann AJ, Walsh TJ, Helfgott D, Holowiecki J, Stockelberg D, Goh YT, Petrini M, Hardalo C, Suresh R, Angulo-Gonzalez D. Posaconazole vs. fluconazole or itraconazole prophylaxis in patients with neutropenia. N Engl J Med. 2007 Jan 25;356(4):348-59. doi: 10.1056/NEJMoa061094. PMID 17251531
- [Background] Pagano L, Verga L, Busca A, Martino B, Mitra ME, Fanci R, Ballanti S, Picardi M, Castagnola C, Cattaneo C, Nadali G, Nosari A, Candoni A, Caira M, Salutari P, Lessi F, Aversa F, Tumbarello M. Systemic antifungal treatment after posaconazole prophylaxis: results from the SEIFEM 2010-C survey. J Antimicrob Chemother. 2014 Nov;69(11):3142-7. doi: 10.1093/jac/dku227. Epub 2014 Jun 19. PMID 24948702
- [Background] Facchinelli D, Marchesini G, Nadali G, Pagano L. Invasive Fungal Infections in Patients with Chronic Lymphoproliferative Disorders in the Era of Target Drugs. Mediterr J Hematol Infect Dis. 2018 Nov 1;10(1):e2018063. doi: 10.4084/MJHID.2018.063. eCollection 2018. PMID 30416695